CLINICAL TRIAL: NCT00104078
Title: Study Evaluating MYO-029 in Adult Muscular Dystrophy
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 3147K2-101
Record Dates: First submitted 2005-02-22; First posted 2005-02-23 (Estimated); Last update posted 2007-12-28 (Estimated); Status verified 2007-12

CONDITIONS: Becker Muscular Dystrophy; Facioscapulohumeral Muscular Dystrophy; Limb-Girdle Muscular Dystrophy
MeSH Terms: conditions — Muscular Dystrophy, Duchenne; Muscular Dystrophy, Facioscapulohumeral; Muscular Dystrophies, Limb-Girdle | interventions — Stamulumab

INTERVENTIONS:
Drug: MYO-029

SUMMARY:
The purpose of this phase I/II, multicenter, safety trial is to study MYO-029 in adult patients with muscular dystrophy.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent.
* Confirmed clinical and molecular diagnosis of Becker Muscular Dystrophy (BMD), Facioscapulohumeral Muscular Dystrophy (FSHD), or Limb-Girdle Muscular Dystrophy (LGMD)
* Independently ambulatory

Exclusion Criteria:

* Patients with certain clinical conditions
* Patients using steroids or other medications with the potential to affect muscle function
* History of sensitivity to monoclonal antibodies or protein pharmaceuticals
* Pregnant or lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108
Dates: Start 2005-02; Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Safety assessment

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, MD, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (9):
- United States (9):
  - Washington D.C., District of Columbia
  - Kansas City, Kansas
  - Baltimore, Maryland
  - Boston, Massachusetts
  - St Louis, Missouri
  - Rochester, New York
  - Columbus, Ohio
  - Dallas, Texas
  - Salt Lake City, Utah